CLINICAL TRIAL: NCT04709094
Title: A Three-Part Phase 1 Study to Evaluate the Potential Drug Interaction Between ACH-0144471 and Warfarin, Bupropion, and Ethinyl Estradiol and Norethindrone (Oral Contraceptive) in Healthy Adult Subjects
Brief Title: A Drug Interaction Study of Danicopan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry); Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-017; CA27858 (Other: Celerion)
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Factor D Inhibitor; Complement; Danicopan; Oral Contraceptive; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — danicopan; Warfarin; Bupropion; ovcon 35; Norinyl

STUDY DESIGN:
Intervention Model Description: Part 1, Part 2, and Part 3 could be conducted concurrently or separately.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Danicopan and Warfarin (Experimental): Period 1: Participants received a single dose of warfarin.
  Period 2: Participants received danicopan three times daily, in addition to coadministration with a single dose of warfarin.
  Scheduled pharmacokinetics (PK) and pharmacodynamics samples were collected, with a washout period of at least 14 days between the dose of warfarin in Period 1 and the first dose of danicopan in Period 2.
  Interventions: Drug: Danicopan; Drug: Warfarin
- Part 2: Danicopan and Bupropion (Experimental): Period 1: Participants received a single dose of bupropion.
  Period 2: Participants received danicopan three times daily, in addition to coadministration with a single dose of bupropion.
  Scheduled PK samples were collected, with a washout period of at least 7 days between the dose of bupropion in Period 1 and the first dose of danicopan in Period 2.
  Interventions: Drug: Danicopan; Drug: Bupropion
- Part 3: Danicopan and EE/NET (Experimental): Period 1: Participants received a single dose of EE/NET.
  Period 2: Participants received danicopan three times daily, in addition to coadministration with a single dose of EE/NET.
  Scheduled PK samples were collected, with a washout period of at least 7 days between the dose of EE/NET in Period 1 and the first dose of danicopan in Period 2.
  Interventions: Drug: Danicopan; Drug: Ethinyl Estradiol/Norethindrone

INTERVENTIONS:
Drug: Danicopan — Danicopan was dosed as 2 x 100 milligram (mg) tablets.
  Other Names: ACH-0144471; ALXN2040
Drug: Warfarin — Warfarin was dosed as 2 x 10 mg and 1 x 5 mg warfarin sodium tablets (Coumadin or generic equivalent).
  Other Names: Coumadin
  Arms: Part 1: Danicopan and Warfarin
Drug: Bupropion — Bupropion was dosed as Wellbutrin (or generic equivalent) as 1 x 100 mg tablet.
  Other Names: Bupropion HCl; Wellbutrin
  Arms: Part 2: Danicopan and Bupropion
Drug: Ethinyl Estradiol/Norethindrone — EE/NET (0.035 mg/1 mg) was dosed as Ortho-Novum-1/35 (or generic equivalent) fixed-dose combination tablets.
  Other Names: Ortho-Novum
  Arms: Part 3: Danicopan and EE/NET

SUMMARY:
This was a 3-part study (Part 1, Part 2, Part 3) with each part being an open-label, fixed sequence, 2-period study in healthy adult participants.

DETAILED DESCRIPTION:
This study was conducted to assess the 2-way interaction between danicopan and warfarin (Part 1), bupropion (Part 2), and ethinyl estradiol/norethindrone (EE/NET) as an oral contraceptive (Part 3).

ELIGIBILITY:
Inclusion Criteria:

1. Parts 1 and 2: adult males or females between 18 and 55 years of age, inclusive, at screening. Part 3: adult females between 18 and 65 years of age, inclusive, at screening.
2. Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at screening.
3. No clinically significant history or presence of electrocardiogram abnormalities at screening.
4. Non-sterile male participants must agree to abstinence or use a highly effective method of contraception.
5. Female participants must be of non-childbearing potential and need not employ a method of contraception.
6. Part 1 only: Participant has a negative fecal occult blood test at screening.

Exclusion Criteria:

1. Clinically significant laboratory abnormalities.
2. History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
3. History or presence of drug or alcohol abuse within previous 2 years, current tobacco/nicotine user, or positive for alcohol and/or drug screen at screening or Day -1 of Period 1.
4. History or presence of clinically significant seizures, head injury, or head trauma.
5. History of procedures that could alter absorption or excretion of orally administered drugs.
6. History of meningococcal infection, or a first-degree relative with a history of meningococcal infection.
7. A history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs.
8. Body temperature ≥ 38.0°Celsius at screening or prior to first dosing in Period 1 or history of febrile illness, or other evidence of infection, within 14 days prior to first dosing.
9. Donation of whole blood from 3 months prior to first dosing, or of plasma from 30 days before first dosing, or receipt of blood products within 6 months prior to first dosing.
10. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days before first dosing, whichever is longer.

    Part 1 Only:
11. History or presence of any of the following, with clinical significance:

    * bleeding disorder(s), including relevant familial history;
    * anemia (for example, history of temporary anemia during pregnancy is acceptable);
    * thromboembolic disease;
    * bleeding in the gastrointestinal tract or central nervous system.
12. Has active severe gingivitis.
13. Clinically significant illness, clinically significant surgery, including tooth extraction, trauma, or head injury, within 28 days before Day 1 of Period 1.
14. Participant is employed or actively involved in any circumstance that would place them at increased risk of hemorrhage during the study (for example, contact sports, strenuous or unaccustomed weight lifting, running, bicycling).
15. Participant has taken large daily doses of vitamin K (> 25 micrograms/daily) and/or has a diet rich in vitamin K 14 days prior to the first dosing.

    Part 2 Only:
16. Any significant finding on the Columbia-suicide severity rating scale.
17. History or presence of any of the following, with clinical significance:

    * bulimia or anorexia nervosa;
    * hypertension;
    * angle-closure glaucoma;
    * seizure disorder;
    * prior seizure to previous bupropion administration;
    * head trauma.

    Part 3 Only:
18. History or presence of:

    * migraines or severe headaches;
    * thrombotic disorders (thrombophlebitis, deep vein thrombosis);
    * cerebrovascular accident;
    * hypertension;
    * transient ischemic attacks;
    * undiagnosed vaginal bleeding;
    * liver tumors or liver disease;
    * jaundice with previous use of oral contraceptives or past pregnancy;
    * diabetes (including gestational diabetes);
    * carcinoma of the endometrium, breast or other known or suspected estrogen dependent neoplasia;
    * family history of first degree relative with breast, ovarian, cervical, or endometrial/uterine cancer;
    * history of abnormal pap smear (high-grade squamous intraepithelial lesion or greater result) including positive human papilloma virus test and/or cervical cancer, or history of cervical procedures including loop electrosurgical excision procedure or conization;
    * any condition that would contraindicate the use of oral contraceptives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-07-28 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Part 1: Area Under The Concentration Versus Time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) Of Single-dose Warfarin Under Multiple Doses Of Danicopan | Up to 168 hours postdose
Part 1: Maximum Observed Concentration (Cmax) Of Single-dose Warfarin Under Multiple Doses Of Danicopan | Up to 168 hours postdose
Part 1: Time To Maximum Observed Concentration (Tmax) Of Single-dose Warfarin Under Multiple Doses Of Danicopan | Up to 168 hours postdose
Part 2: AUC0-inf Of Single-dose Bupropion Under Multiple Doses Of Danicopan | Up to 96 hours postdose
Part 2: Cmax Of Single-dose Bupropion Under Multiple Doses Of Danicopan | Up to 96 hours postdose
Part 2: Tmax Of Single-dose Bupropion Under Multiple Doses Of Danicopan | Up to 96 hours postdose
Part 3: AUC0-inf Of Single-dose EE/NET Under Multiple Doses Of Danicopan | Up to 96 hours postdose
Part 3: Cmax Of Single-dose EE/NET Under Multiple Doses Of Danicopan | Up to 96 hours postdose
Part 3: Tmax Of Single-dose EE/NET Under Multiple Doses Of Danicopan | Up to 96 hours postdose

SECONDARY OUTCOMES:
Part 1: International Normalized Ratio (INR) Of Single-dose Warfarin Under Multiple Doses Of Danicopan | Up to 168 hours postdose
  Blood samples will be collected for prothrombin time/INR determination.
Part 1: Number Of Participants With Treatment-emergent Adverse Events (TEAEs) After Multiple Doses Of Danicopan Coadministered With A Single Dose Of Warfarin | Day 1 (postdose) through follow-up (14 [+/- 2] days after last study drug administration)
Part 2: Number Of Participants With TEAEs After Multiple Doses Of Danicopan Coadministered With A Single Dose Of Bupropion | Day 1 (postdose) through follow-up (14 [+/- 2] days after last study drug administration)
Part 3: Number Of Participants With TEAEs After Multiple Doses Of Danicopan Coadministered With A Single Dose Of EE/NET | Day 1 (postdose) through follow-up (14 [+/- 2] days after last study drug administration)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Study Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No